CLINICAL TRIAL: NCT02718495
Title: A Phase I/II, Multi-center, Randomized, Placebo-Controlled, Study Designed to Assess the Safety, Tolerability, and Pharmacokinetics of PTI-428 in Subjects With Cystic Fibrosis
Brief Title: Study Assessing PTI-428 Safety, Tolerability, and Pharmacokinetics in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Proteostasis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTI-428-01
Record Dates: First submitted 2016-03-10; First posted 2016-03-24 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part A (Placebo Comparator): Part A consists of two treatment groups, SAD and MAD. Both treatment groups will consist of 3 cohorts. In SAD, subjects will receive a single dose of PTI-428 or placebo. In MAD, subjects will receive once daily dosing of PTI-428 or placebo for 7 days.
  Interventions: Drug: PTI-428; Drug: Placebo
- Part B (Placebo Comparator): Part B will consist of 2 cohorts. Subjects will receive once daily dosing of PTI-428 or placebo for 28 days.
  Interventions: Drug: PTI-428; Drug: Placebo
- Part C (Placebo Comparator): Part C will consist of 3 cohorts. Subjects will receive once daily dosing of PTI-428 or placebo for 28 days.
  Interventions: Drug: PTI-428; Drug: Placebo

INTERVENTIONS:
Drug: PTI-428
Drug: Placebo

SUMMARY:
This trial will consist of three arms: Part A, Part B, and Part C. Part A has two groups. The first group will enroll adult subjects with cystic fibrosis (CF) into a single ascending dose (SAD) treatment group. The second group will enroll adult subjects with CF, including those on background treatment with ORKAMBI® and those not on a cystic fibrosis transmembrane conductance regulator (CFTR) modulator, into a multiple ascending dose (MAD) treatment group. Part B will enroll adult subjects with CF currently on stable ORKAMBI® background therapy for a minimum of 3 months into a Phase II treatment group consisting of two cohorts. Part C will enroll adult subjects with CF, including those on background treatment with KALYDECO® and those not on a CFTR modulator, into a Phase II treatment group consisting of three cohorts. Approximately 136 subjects will be enrolled.

DETAILED DESCRIPTION:
PART A The SAD treatment group is comprised of 3 cohorts where subjects will be randomized to either PTI-428 or placebo. Following the conclusion of at least 3 SAD treatment groups, a set of adult subjects diagnosed with CF will participate in an assigned MAD treatment group. The MAD treatment group is comprised of 3 cohorts. MAD Cohort 1 will enroll adult subjects with CF currently on stable ORKAMBI® background therapy for a minimum of 3 months at the time of randomization. MAD Cohorts 2 and 3 will enroll adult subjects with CF who are not currently on any background therapies. Subjects in all MAD cohorts will be randomized to either PTI-428 or placebo. Each dose will be administered once daily (QD) for a total of 7 Days.

PART B Following the conclusion of MAD Cohort 1, a set of adult subjects diagnosed with CF currently on stable ORKAMBI® background therapy for a minimum of 3 months will participate in Part B. The Part B Phase II treatment group is comprised of 2 cohorts where subjects will be randomized to either PTI-428 or placebo. Each dose will be administered QD for a total of 28 days.

PART C Following the conclusion of Part B Phase II, a set of adult subjects diagnosed with CF will participate in Part C. The Part C Phase II treatment group is comprised of 3 cohorts. Part C Cohort 1 will enroll adult subjects with CF who are eligible to take, but not currently taking, ORKAMBI® in accordance with the approved label. Part C Cohort 2 will enroll adult subjects with CF currently on stable KALYDECO® background therapy for a minimum of 3 months at the time of randomization. Part C Cohort 3 will enroll adult subjects with CF who are not currently on any background therapies and are pancreatic sufficient. Each PTI-428 or placebo dose will be administered QD for a total of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF.
* Forced expiratory volume in 1 second (FEV1) 40-90% predicted.
* Non-smoker and non-tobacco user for a minimum of 30 days prior to screening and for the duration of the study.

Exclusion Criteria:

* Participation in another clinical trial or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, prior to Study Day 1.
* History of cancer within the past five years (excluding cervical CIS with curative therapy for at least one year prior to screening and non-melanoma skin cancer).
* History of organ transplantation.
* Any sinopulmonary infection or CF exacerbation requiring a change or addition of medication (including antibiotics) within 1 month of Study Day 1 or any other clinically significant infection as determined by the investigator within 1 month of Day 1.
* History of alcohol or drug abuse or dependence within 12 months of screening as determined by the Investigator.
* Male and female of child-bearing potential, unless they are using highly effective methods of contraception during participation in the clinical study and for 4 weeks after termination from study.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
SAD: safety and tolerability as assessed by adverse events, safety labs: hematology, chemistry, and urinalysis, electrocardiograms (ECGs), physical examinations, and vital signs | Baseline to Day 7
MAD: safety and tolerability as assessed by adverse events, pulomonary function tests, safety labs: hematology, chemistry, and urinalysis, electrocardiograms (ECGs), physical examinations, and vital signs | Baseline to Day 14
Part B and Part C Cohorts 2 and 3: safety and tolerability as assessed by adverse events, safety labs: hematology, chemistry, and urinalysis, electrocardiograms (ECGs), physical examinations, and vital signs | Baseline to Day 35
Part C Cohort 1: safety and tolerability as assessed by adverse events, safety labs: hematology, chemistry, and urinalysis, electrocardiograms (ECGs), physical examinations, and vital signs | Baseline to Day 49

SECONDARY OUTCOMES:
SAD: apparent terminal half-life (t1/2) of single oral dose | Baseline through 72 hours post dose
SAD: time to reach maximum plasma concentration (Tmax) of single oral dose | Baseline through 72 hours post dose
SAD: maximum plasma concentration (Cmax) of single oral dose | Baseline through 72 hours post dose
SAD: area under the concentration-time curve from time 0 to time of last measurable concentration (AUC0-t) of single oral dose | Baseline through 72 hours post dose
MAD: t1/2 of multiple oral doses | Baseline through 24 hours post Day 7 dose
MAD: Tmax of multiple oral doses | Baseline through 24 hours post Day 7 dose
MAD: Cmax of multiple oral doses | Baseline through 24 hours post Day 7 dose
MAD: AUC0-t of multiple oral doses | Baseline through 24 hours post Day 7 dose
MAD: area under the concentration-time curve from time 0 to infinity (AUC0-∞) of multiple oral doses | Baseline through 24 hours post Day 7 dose
Part B and Part C Cohorts 2 and 3: t1/2 of multiple oral doses | Baseline through 24 hours post Day 28 dose
Part B and Part C Cohorts 2 and 3: Tmax of multiple oral doses | Baseline through 24 hours post Day 28 dose
Part B and Part C Cohorts 2 and 3: Cmax of multiple oral doses | Baseline through 24 hours post Day 28 dose
Part B and Part C Cohorts 2 and 3: AUC0-t of multiple oral doses | Baseline through 24 hours post Day 28 dose
Part B and Part C Cohorts 2 and 3: AUC0-∞ of multiple oral doses | Baseline through 24 hours post Day 28 dose
Part B and Part C Cohorts 2 and 3: change in forced expiratory volume in one second (FEV1) over time | Baseline through Day 35
Part B and Part C Cohorts 2 and 3: change in sweat chloride over time | Baseline through Day 35
Part B and Part C Cohorts 2 and 3: change in weight over time | Baseline through Day 35
Part C Cohort 1: t1/2 of multiple oral doses | Baseline through Day 42
Part C Cohort 1: Tmax of multiple oral doses | Baseline through Day 42
Part C Cohort 1: Cmax of multiple oral doses | Baseline through Day 42
Part C Cohort 1: AUC0-t of multiple oral doses | Baseline through Day 42
Part C Cohort 1: AUC0-∞ of multiple oral doses | Baseline through Day 42
Part C Cohort 1: change in FEV1 over time | Baseline through Day 49
Part C Cohort 1: change in sweat chloride over time | Baseline through Day 49
Part C Cohort 1: change in weight over time | Baseline through Day 49

OTHER OUTCOMES:
SAD: change in nasal epithelial CFTR mRNA and protein expression | Baseline through Day 7
MAD: change in nasal epithelial CFTR mRNA and protein expression | Baseline through Day 14
MAD: change in sweat chloride over time | Baseline through Day 14
Part B and Part C Cohorts 2 and 3: change in nasal epithelial CFTR mRNA and protein expression | Baseline through Day 35
Part B and Part C Cohorts 2 and 3: change in CFQ-R over time | Baseline through Day 28
Part C Cohort 1: change in nasal epithelial CFTR mRNA and protein expression | Baseline through Day 49
Part C Cohort 1: change in CFQ-R over time | Baseline through Day 42
Part C Cohort 3: change in fecal elastase over time | Baseline through Day 35
Part C Cohort 3: change in fecal calprotectin over time | Baseline through Day 35

CONTACTS AND LOCATIONS:
Locations (29):
- United States (20):
  - Stanford University Medical Center, Stanford, California
  - Central Florida Pulmonary Group, Altamonte Springs, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - St. Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Northwestern University Memorial Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Quintiles Overland Park Phase 1 Unit, Overland Park, Kansas
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Childrens Hospital Boston, Boston, Massachusetts
  - Universiy of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Lung Specialists, Las Vegas, Nevada
  - Duke University Health System, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (4):
  - St. Paul's Hospital Pacific Lung Research Center, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Recherches Cliniques de Montreal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
- University of Copenhagen Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Groupe Hospitalier Pellegrin - Hôpital des Enfants, Bordeaux
  - Hôpital Cochin, Paris
- Germany (2):
  - Charite - Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Frankfurt-Zentrum der Inneren Medizin, Frankfurt

IPD SHARING:
Plan to Share IPD: Yes